CLINICAL TRIAL: NCT05797064
Title: Establishment of a Feasibility Model for Predicting Natural Orifice Specimen Extraction Surgery (NOSES) Based on Machine Learning.
Brief Title: Establishment of a Feasibility Model for NOSE Surgery Based on Machine Learning
Status: Not yet recruiting | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanxin Luo,MD, Principal Investigator, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: 1010PY(2022)-09
Record Dates: First submitted 2023-03-21; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Machine Learning; Surgery; Rectosigmoid Cancer; Natural Orifice Specimen Extraction Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training set: The training set is a dataset used to train the model, which includes randomly enrolled patients with colon and rectal cancer. The inputs include data such as gender, age, height, weight, BMI, tumor stage, tumor pathology type, and the output information is whether NOSES surgery was successful or not. During training, the model learns from this dataset to make predictions on whether new patients with colon and rectal cancer can undergo NOSES surgery successfully.
  Interventions: Procedure: Natural Orifice Specimen Extraction Surgery
- test set: The test set is a dataset used to evaluate the performance of a trained machine learning model. It includes another randomly enrolled group of patients with colon and rectal cancer, as well as their clinical and pathological data and surgical outcomes. The outputs are not used during training, but are used to test the trained model to evaluate its predictive ability on unknown data. The purpose is to evaluate the model's generalization ability, that is, its performance on new and unknown data.
  Interventions: Procedure: Natural Orifice Specimen Extraction Surgery

INTERVENTIONS:
Procedure: Natural Orifice Specimen Extraction Surgery — Natural Orifice Specimen Extraction Surgery (NOSES) is a minimally invasive surgical technique that aims to reduce the size and number of incisions required during certain surgeries. In NOSES, the surgical specimen (such as a diseased organ or tumor) is removed from the body through a natural orifice (such as the mouth, anus, or vagina), rather than through an incision in the abdominal wall. In this trial, we will extract surgical specimens from the rectum to reduce trauma to the abdominal wall.
  Other Names: NOSES

SUMMARY:
The goal of this observational study is to test in patients with resectable rectosigmoid cancers. The main question it aims to answer is establishment of a feasibility model for predicting natural orifice specimen extraction surgery (NOSES) based on machine learning.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with colorectal cancer or large adenoma who are suitable for laparoscopic colorectal surgery;
2. Tumor staging ≤ T3 without invasion of surrounding organs;
3. No abdominal seeding or distant organ metastasis;
4. Clear and complete imaging data (CT, pelvic MRI) that can be processed by a computer;
5. Feasible evaluation and determination for obtaining specimens through the rectal channel during preoperative and intraoperative assessments.

Exclusion Criteria:

1. Contraindications for laparoscopic colorectal surgery;
2. Tumor staging is T4, or there are cancer nodules;
3. Presence of metastasis or distant organ metastasis;
4. Incomplete imaging data;
5. Preoperative intestinal obstruction;
6. Tumor or specimen diameter larger than the transverse diameter of the pelvic outlet;
7. Previous rectal radiotherapy;
8. Unsuitable evaluation and determination for obtaining specimens through the rectal channel during preoperative and intraoperative assessments.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with resectable rectosigmoid cancer.
Sampling Method: Non-Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The number of successful operations performed | 3 years
  Accuracy will be calculated by the number of successful operations performed
The number of successful operations actually completed. | 3 years
  Accuracy will be calculated by the number of successful operations actually completed.

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliate Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided